CLINICAL TRIAL: NCT00919815
Title: A Randomised Double Blind Controlled Trial Comparing Ciclosporin and Prednisolone in the Treatment of New Leprosy Type 1 Reactions
Brief Title: Ciclosporin in the Management of New Type 1 Reactions in Leprosy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Homes and Hospitals of St Giles (Other); Alert Hospital, Ethiopia (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Saba Lambert, Clinical Research Fellow, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITCRBY24-T1RA
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Leprosy
Keywords: Leprosy; Type 1 Reactions; Prednisolone; Ciclosporin
MeSH Terms: conditions — Leprosy | interventions — Cyclosporine; Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ciclosporin arm (Experimental): ciclosporin reducing regimen lasting 24 weeks (additional prednisolone given for the first four weeks)
  Interventions: Drug: Ciclosporin
- prednisolone (Active Comparator): standard course of prednisolone given in a reducing regimen over 24 weeks
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Ciclosporin — Ciclosporin 7.5mg/kg - reducing regimen over 24 weeks (additional prednisolone given for the first four weeks)
  Other Names: Cyclosporine; Cyclosporine A
  Arms: ciclosporin arm
Drug: Prednisolone — prednisolone 40mg daily then reducing regimen over 24 weeks
  Other Names: corticosteroids
  Arms: prednisolone

SUMMARY:
Study 1A: Ciclosporin in the management of new Type 1 Reactions in Leprosy

Objective: A randomised double blind controlled trial comparing Ciclosporin and Prednisolone,to determine whether treatment with Ciclosporin gives the same outcome in the treatment of new Type 1 Reactions as Prednisolone.

DETAILED DESCRIPTION:
We tested our hypothesis that ciclosporin would be as effective as prednisolone in the treatment of patients with leprosy reactions and nerve function impairment and that patients treated with ciclosporin would have fewer side effects than patients treated with prednisolone. A randomised controlled trial comparing ciclosporin and prednisolone in the treatment of acute leprosy T1R was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical evidence of T1R with new nerve function impairment (NFI).
* Aged 18-65
* Weigh more than 30Kg

Exclusion Criteria:

* Unwillingness to give informed consent
* Patients with severe active infections such as tuberculosis
* Pregnant or breastfeeding women (see Appendix II)
* Those with renal failure, abnormal renal function, hypertensive
* Patients taking thalidomide currently or within the last 3 months
* Patients not willing to return for follow-up
* Women of reproductive age not willing to use contraception for the duration of the study ( see Appendix II)
* HIV positive patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
improvement in nerve function and Clinical Severity Score | at week 4, 20, 28

SECONDARY OUTCOMES:
Incidence of adverse events | up to 36 weeks
Number of T1R recurrence episodes per patient in each treatment arm | up to 36 weeks
Severity of T1R recurrence for patients in each treatment arm | up to 36 weeks
extra prednisolone needed to control reaction | up to 36 weeks
6. Difference in score in Quality of Life assessment between start and end of treatment for patients in each treatment arm | 36 weeks
Mean time to recurrence of T1R for patients in each treatment arm | up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana Lockwood, MBChB, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Alert Hospital, Addis Ababa, Ethiopia